CLINICAL TRIAL: NCT03558854
Title: Evaluation of Effectiveness of Acetylsalicylic Acid on Markers of Vascular Dysfunction in Patients With Systemic Sclerosis
Brief Title: Evaluation of Effectiveness of Acetylsalicylic Acid on Markers of Vascular Dysfunction in Scleroderma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Cristiane Kayser, Principal investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0246/2018
Record Dates: First submitted 2018-05-03; First posted 2018-06-15 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Acetylsalicylic acid; Vascular dysfunction
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASA group (Active Comparator): Pill containing 100 mg of acetylsalicylic acid, taken once daily for 04 weeks
  Interventions: Drug: Acetylsalicylic acid
- Placebo oral capsule group (Placebo Comparator): Identical pill containing placebo, taken once daily for 04 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Acetylsalicylic acid — Patients will be randomized to take one pill of either acetylsalicylic acid or placebo once daily for 4 weeks
  Arms: ASA group
Drug: Placebo oral capsule — Patients will be randomized to take one pill of either acetylsalicylic acid or placebo once daily for 4 weeks
  Arms: Placebo oral capsule group

SUMMARY:
Systemic sclerosis is a chronic autoimmune disease characterized by vascular changes in the microcirculation (small blood vessels) and progressive fibrosis of the skin and internal organs. It is believed that vascular changes, expressed early by the Raynaud phenomenon, precede fibrosis and organic dysfunction. There is no available treatment that reverses the vascular damage caused by the disease to the moment, although there are several medications recommended for the relief of manifestations due to vascular injury. Acetylsalicylic acid (ASA) is one of the medications that can be used for the treatment of vascular injury present in systemic sclerosis, but still without a fully proven benefit. This study aims to evaluate the effectiveness of ASA on microcirculation alterations in patients with systemic sclerosis by performing three exams: periungual panoramic capillary microscopy, videocapillaroscopy and laser Doppler imaging. In addition, a blood sample will be collected for dosing the following vascular lesion markers: endothelin-1, von Willebrand factor, thromboxane, and platelet-derived, endothelial-derived and monocyte-derived microparticles.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill Systemic sclerosis EULAR/American College of Rheumatology 2013 classification criteria;
* Pharmacological treatment with stable dosages for the last three months.

Exclusion Criteria:

* Pregnancy;
* Use of anticoagulants, NSAIDs or antiplatelets drugs;
* Diagnose of other autoimmune rheumatic diseases, coronary diseases, cerebrovascular diseases and severe peripheral artery diseases;
* Active infection;
* Contraindication to acetylsalicylic acid use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Serum level of thromboxane B2 | Baseline and 4 weeks
  Measured by ELISA

SECONDARY OUTCOMES:
Serum level of platelet-derived, endothelial-derived and monocyte-derived microparticles | Baseline and 4 weeks
  Measured by flow cytometry
Serum level of von Willebrand factor | Baseline and 4 weeks
  Measured by ELISA
Serum level of endothelin-1 | Baseline and 4 weeks
  Measured by ELISA
Digital blood flow | Baseline and 4 weeks
  Measured by laser Doppler imaging

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Kayser, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Systemic Sclerosis Outpatient Clinic, Hospital São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Under discussion